CLINICAL TRIAL: NCT06549569
Title: Tilapia Fish Skin Coverage in Acute Thermal Burn; Experimental and Histopathological Study
Brief Title: Burn Coverage of Burn by Tilapia Fish Skin
Acronym: TFS
Status: Completed | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Amira Anter, resident, Aswan University
Other Study IDs: 696/11/22
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Tilapia Fish Skin in Burn Coverage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TFS: thermal burn coverage with Tilapia fish skin
  Interventions: Procedure: TFS
- regular dressing: thermal burn coverage with regular dressing
  Interventions: Procedure: TFS

INTERVENTIONS:
Procedure: TFS — burn coverage with TFS

SUMMARY:
The goal of this experimental study is to compare TFS and regular dressings as coverage for acute thermal burns. The main question it aims to answer is:

Is TFS effective in treating thermal burns? burn induction was done on rabbits to obtain second-degree thermal burn, followed by coverage with TFS

DETAILED DESCRIPTION:
Nile Tilapia Fish Skin (NTFS) has been suggested as an option for biological material for the management of burns. Nile Tilapia Fish Skin also presented a large composition of type I collagen, morphology similar to human skin and high resistance and tensile extension at the break. We chose Baladi rabbits for their relatively ease of handling, accommodation and resistance to surgical aggressions and infectious processes, with low mortality. However, the choice of male rabbits is due to variations in hormonal cycles in females that could intervene in the process of tissue repair.

This experimental model was established to evaluate healing process and outcome results after application of Tilapia Fish Skin on acute contact thermal that was done in order to obtain injuries with the same size and depth.

ELIGIBILITY:
Inclusion Criteria:

- healthy male one year old rabbit

Exclusion Criteria:

* female unhealthy rabbits

Ages: 1 Year to 18 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: animal rabbits
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Tilapia Fish Skin Coverage in Acute Thermal Burn | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Anter, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No